CLINICAL TRIAL: NCT02049515
Title: A Study of IPI-145 and Ofatumumab in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Previously Enrolled in Study IPI-145-07 Duvelisib (IPI-145)
Brief Title: A Phase 3 Extension Study of Duvelisib and Ofatumumab in Participants With CLL/SLL Previously Enrolled in Study IPI-145-07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-12; 2013-003639-31 (EudraCT Number)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Phase 3; CLL/SLL; PI3K
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPI-145 (Experimental): IPI-145 was administered orally and supplied as 5 mg and 25 mg formulated capsules.
  Interventions: Drug: IPI-145
- Ofatumumab (Active Comparator): Ofatumumab was administered as an intravenous (IV) infusion and was supplied in single-use vials at two strengths, 100 mg/5 milliliters (mL) and 1000 mg/50 mL.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: IPI-145 — PI3K Inhibitor
  Other Names: Duvelisib; Copiktra; PI3K Inhibitor
  Arms: IPI-145
Drug: Ofatumumab — Monoclonal antibody
  Other Names: Arzerra
  Arms: Ofatumumab

SUMMARY:
A Phase 3 (extension) clinical trial to examine the efficacy of IPI-145 (duvelisib) monotherapy or ofatumumab monotherapy in participants with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who experienced disease progression after treatment with IPI-145 or ofatumumab in study IPI-145-07 (NCT02004522).

DETAILED DESCRIPTION:
The study was designed as an open-label, two-arm extension evaluation to enable participants who experienced radiologically confirmed disease progression in study IPI-145-07 to receive the alternative treatment (either IPI-145 or ofatumumab) other than what was received during study IPI-145-07.

Participants who previously had received ofatumumab in study IPI-145-07 received a starting dose of 25 milligrams (mg) IPI-145 twice daily continuously in a 21-day cycle for Cycle 1, followed by 28-day treatment cycles thereafter for up to 11 cycles or until disease progression, discontinuation from study participation, or start of subsequent therapy, whichever occurred first. After completing approximately 11 cycles of treatment with duvelisib, participants who, in the judgment of the investigator, may have derived benefit from continued treatment may have continued to receive additional cycles of duvelisib until disease progression or unacceptable toxicity. However, to receive additional cycles of duvelisib beyond 11 cycles, participants must have had evidence of response and CLL/SLL requiring treatment according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL)/International Working Group by Cycle 12 Day 1.

Participants who previously received IPI-145 in study IPI-145-07 received treatment consistent approved product labeling which consisted of a starting dose of 300 mg ofatumumab on Day 1, followed by seven weekly doses of 2000 mg. Thereafter, participants received 2000 mg ofatumumab once every month for four months unless disease progression or unacceptable toxicity occurred. Administration of ofatumumab was not to exceed the 12 doses (within 7 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Received either IPI-145 or ofatumumab while participating in study IPI-145-07 and experienced radiologically confirmed disease progression
* Diagnosis of active CLL or SLL that met at least one of the IWCLL 2008 criteria for requiring treatment
* Measurable disease with a lymph node or tumor mass >1.5 centimeters in at least one dimension as assessed by computed tomography (CT)
* Eastern Cooperative Oncology Group performance status of 0-2
* Must have met the following laboratory parameters:

  1. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤3 x upper limit of normal (ULN)
  2. Total bilirubin ≤1.5 x ULN
  3. Serum creatinine ≤2.0 x ULN
  4. Hemoglobin ≥8.0 grams/deciliter (g/dL) with or without transfusion support
  5. Platelet count ≥10,000 microliters (μL) with or without transfusion support
* For women of childbearing potential (WCBP): negative serum β-human chorionic gonadotropin pregnancy test within one week before first dose (WCBP defined as a sexually mature woman who had not undergone surgical sterilization or who had not been naturally post-menopausal for at least 24 consecutive months [women ≤55 years] or 12 consecutive months [women >55 years])
* Willingness of male and female participants who were not surgically sterile or postmenopausal to use medically acceptable methods of birth control from the first dose of study drug to 30 days after the last dose of duvelisib and for 12 months after last dose of ofatumumab. Sexually active men, and women using oral contraceptive pills, should also have used barrier contraception
* Ability to voluntarily sign consent for and adhere to the entire study visit schedule and all protocol requirements
* Signed and dated institutional review board/independent ethics committee-approved informed consent form before any study-specific screening procedures are performed

Exclusion Criteria:

* Discontinued study participation in Verastem-sponsored IPI-145-07 study
* Greater than 3 months from confirmed progressive disease on Study IPI-145-07
* History of Richter's transformation or prolymphocytic leukemia
* Autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura that was uncontrolled or requires >20 mg daily of prednisone (or equivalent) to maintain hemoglobin >8.0 g/dL or platelets >10,000 μL without transfusion support
* Known central nervous system (CNS) lymphoma or leukemia; participants with symptoms of CNS disease must have had a negative CT scan or negative diagnostic lumbar puncture prior to first dose
* Use of any anticancer medication from documented progressive disease on Study IPI-145-07 to enrollment (Note: corticosteroids to manage CLL/SLL-related symptoms were allowed)
* Ongoing systemic bacterial, fungal, or viral infections at the time of initiation of study treatment (defined as requiring IV antimicrobial, antifungal or antiviral agents) (Participants on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met and there is no evidence of active infection at Screening and/or Cycle 1 Day 1 [predose])
* Human immunodeficiency virus infection
* Prior, current, or chronic hepatitis B or hepatitis C infection
* History of alcohol abuse or chronic liver disease (other than metastatic disease to the liver)
* Unable to receive prophylactic treatment for pneumocystis and herpes simplex virus
* Baseline QT interval corrected with Fridericia's method >480 milliseconds Note: this criterion did not apply to participants with a right or left bundle branch block
* Concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix, bladder, or prostate not requiring treatment. Participants with previous malignancies were eligible provided that they had been disease-free for ≥2 years
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Unstable or severe uncontrolled medical condition (for example, unstable cardiac function, unstable pulmonary condition), or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, have increased the participant's risk while participating in this study
* Prior surgery or gastrointestinal dysfunction that may have affected drug absorption (for example, gastric bypass surgery, gastrectomy)
* Participants to receive duvelisib: Administration of medications or foods that were strong inhibitors or inducers of cytochrome P450 3A within 2 weeks of starting duvelisib
* Major surgery or invasive intervention within 4 weeks prior to first dose
* Pregnant or breastfeeding women
* Participants to receive ofatumumab: hypersensitivity to ofatumumab or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-12; Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (60):
- United States (12):
  - La Jolla, California
  - Denver, Colorado
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Boston, Massachusetts
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Charlottesville, Virginia
- Australia (3):
  - Bedford Park
  - East Melbourne
  - Melbourne
- Austria (3):
  - Linz
  - Vienna
  - Wels
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Sint-Niklaas
- France (10):
  - Argenteuil
  - Bobigny
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - La Roche-sur-Yon
  - Limoges
  - Nantes
  - Rennes
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Berlin
  - Leer
  - Ulm
- Hungary (6):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Pécs
  - Szeged
- Italy (8):
  - Catania
  - Lecce
  - Meldola
  - Milan
  - Padua
  - Ravenna
  - Rimini
  - Roma
- New Zealand (2):
  - Auckland
  - Palmerston North
- Spain (3):
  - Barcelona
  - Madrid
  - Pamplona
- United Kingdom (6):
  - Bournemouth
  - Leeds
  - Manchester
  - Nottingham
  - Oxford
  - Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants previously enrolled in study IPI-145-07 (NCT02004522) who experienced radiologically confirmed disease progression while on treatment in that study were eligible to participate in this study.
Groups:
- IPI-145: IPI-145 was administered orally and supplied as 5 milligram (mg) and 25 mg formulated capsules.
Period: Overall Study
Arm/Group | IPI-145 | Ofatumumab
Started | 90 | 9
Received at Least 1 Dose of Study Drug (All-treated analysis set: all participants who received any amount of study drug (IPI-145 or ofatumumab).) | 90 | 9
Completed | 0 | 3
Not Completed | 90 | 6
Not completed — Adverse Event | 46 | 2
Not completed — Protocol-specified Disease Progression | 23 | 2
Not completed — Death | 6 | 0
Not completed — Physician Decision | 5 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Termination of the Study by Sponsor | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Clinical Deterioration | 1 | 0
Not completed — Need Treatment for Metastatic Melanoma | 1 | 0
Not completed — Treatment Interruption >42 Days | 1 | 0
Not completed — Suspected and Unconfirmed Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: All-treated analysis set: all participants who received any amount of study drug (IPI-145 or ofatumumab).
Groups:
- Ofatumumab: Ofatumumab was administered as an IV infusion and was supplied in single-use vials at two strengths, 100 mg/5 mL and 1000 mg/50 mL.
- Total: Total of all reporting groups
Arm/Group | IPI-145 | Ofatumumab | Total
Number analyzed (Participants) | 90 | 9 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 3 | 38
  >=65 years | 55 | 6 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 4 | 37
  Male | 57 | 5 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 82 | 9 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best response (per investigator assessment) of complete response (CR), CR with incomplete marrow recovery (CRi), partial response (PR), or PR with lymphocytosis (PRwL), according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) or revised International Working Group Response (IWG) Criteria, with modification for treatment-related lymphocytosis. The 95% confidence interval was calculated using exact binomial method. Select IWCLL criteria for tumor load assessed by computed tomography (CT): CR/CRi (CLL only), lymphadenopathy (none >1.5 centimeters [cm]), hepatomegaly/splenomegaly (none); PR, lymphadenopathy/hepatomegaly/splenomegaly (decrease ≥50%); PRwL, lymphadenopathy only (decrease ≥50%). Select IWG criteria for tumor load assessed by CT: CR, lymphadenopathy/hepatomegaly/splenomegaly (normal size); PR, lymphadenopathy/hepatomegaly/splenomegaly (decrease ≥50%); PRwL, lymphadenopathy only (decrease ≥50%).
Time Frame: Until progressive disease (PD), death, or other anticancer therapy is initiated (up to 4.5 years)
Population: All-treated analysis set: all participants who received any amount of study drug (IPI-145 or ofatumumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IPI-145 | Ofatumumab
Number analyzed (Participants) | 90 | 9
percentage of participants | 76.7 [66.6 to 84.9] | 0 [0 to 0]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of response per investigator assessment to either PD or death due to any cause. DOR was evaluated using the Kaplan-Meier method based on all treated participants with a documentation of response (that is, CR, CRi, PR, or PRwL) as determined by investigator assessment. Select IWCLL criteria for tumor load assessed by CT: CR/CRi (CLL only), lymphadenopathy (none >1.5 cm), hepatomegaly/splenomegaly (none); PR, lymphadenopathy/hepatomegaly/splenomegaly (decrease ≥50%); PRwL, lymphadenopathy only (decrease ≥50%). Select IWG criteria for tumor load assessed by CT: CR, lymphadenopathy/hepatomegaly/splenomegaly (normal size); PR, lymphadenopathy/hepatomegaly/splenomegaly (decrease ≥50%); PRwL, lymphadenopathy only (decrease ≥50%).
Time Frame: From the first documentation of response to the first documentation of PD or death due to any cause (up to 4.5 years)
Population: All-treated analysis set: all participants who received any amount of study drug (IPI-145 or ofatumumab). DOR was evaluated using the Kaplan-Meier method based on all treated participants with documentation of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IPI-145 | Ofatumumab
Number analyzed (Participants) | 90 | 0
months | 14.9 [8.55 to 18.6] |

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose of study treatment to the first documentation of either investigator-assessed PD or death resulting from any cause. PFS was determined using the Kaplan-Meier method based on all treated participants with a documentation of response (that is, CR, CRi, PR, or PRwL) as determined by investigator assessment.
Time Frame: From the first dose of study treatment to the first documentation of PD or death from any cause (up to 4.5 years)
Population: All-treated analysis set: all participants who received any amount of study drug (IPI-145 or ofatumumab). PFS was determined using the Kaplan-Meier method based on all treated participants with documentation of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IPI-145 | Ofatumumab
Number analyzed (Participants) | 90 | 0
months | 15.3 [12.2 to 20.6] |

ADVERSE EVENTS:
Time Frame: 4.5 years
Arm/Group | IPI-145 | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 20/90 | 2/9
Serious Adverse Events (participants affected / at risk) | 68/90 | 4/9
Other Adverse Events (participants affected / at risk) | 80/90 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPI-145 (N=90) | Ofatumumab (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 1
Colitis (Gastrointestinal disorders) | 8 | 0
Pyrexia (General disorders) | 3 | 0
Disease progression (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Drug intolerance (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0
Pseudomonal sepsis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 13 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis lichenoides et varioliformis acuta (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arterial rupture (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IPI-145 (N=90) | Ofatumumab (N=9)
Neutropenia (Blood and lymphatic system disorders) | 23 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 1
Anaemia (Blood and lymphatic system disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 43 | 0
Vomiting (Gastrointestinal disorders) | 10 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 0
Nausea (Gastrointestinal disorders) | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Pyrexia (General disorders) | 21 | 0
Asthenia (General disorders) | 11 | 0
Oedema peripheral (General disorders) | 6 | 0
Bronchitis (Infections and infestations) | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 6 | 1
Lipase increased (Investigations) | 9 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0
Headache (Nervous system disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Rash (Skin and subcutaneous tissue disorders) | 21 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/33 | 1/4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/33 | 1/4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Weight decreased (Investigations) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02049515/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02049515/SAP_001.pdf